CLINICAL TRIAL: NCT04228653
Title: A Long-Term Follow-up Safety Study for Patients With Idiopathic Parkinson's Disease (PD) Implanted With the DDS and/or Who Received Treatment in the Main Study and/or Extension Study
Brief Title: Long-Term Follow-up Safety After DDS Implantation With/Without CDNF Infusions
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Renishaw (Industry)
Collaborators: Herantis Pharma Plc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-CD-CL-2004
Record Dates: First submitted 2019-08-21; First posted 2020-01-14 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease; Movement Disorders; Neuro-Degenerative Disease; Nervous System Diseases; Brain Diseases
Keywords: Parkinson; CDNF; Drug Delivery System; Intracerebral; Parkinson Disease; Nervous System Disease; Movement Disorders; Brain Diseases; Neurodegenerative Diseases; Parkinsonian Disorders; Basal Ganglia Diseases; Central Nervous System Diseases; Dopamine; Cardiotonic Agents; Sympathomimetrics; Autonomic Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Dopamine Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action; Protective Agents
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Nervous System Diseases; Brain Diseases; Neurodegenerative Diseases; Parkinsonian Disorders; Basal Ganglia Diseases; Central Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No Arm (Experimental): As this is the follow up study, there are no arms
  Interventions: Device: Renishaw Drug Delivery System

INTERVENTIONS:
Device: Renishaw Drug Delivery System — Device that allows pharmaceuticals to be delivered into the brain is to be assessed over a period of time to inform of the long term safety of the implanted device.

SUMMARY:
This study is a follow up to the HP-CD-CL-2002 clinical study. It evaluates the long-term safety in patients with Parkinson's disease after implantation of an investigational drug delivery system (DDS) with or without infusions of CDNF. All patients will have at least the port explanted.

DETAILED DESCRIPTION:
A patients participation in the study will last for up to 4 years and will include up to nine visits:

* Screening (1 visit, same as HP-CD-CL-2003 End-of-Study visit)
* Pre-surgery / explantation surgery / post-surgery (3 visits)
* Safety (4 visits)
* DAT-PET (Dopamine Transporter - Positron Emission Tomography) examination (1 visit)
* End-of-study visit (1 visit)

Study examinations and assessments:

* Physical examination: pulse rate, blood pressure, temperature, body weight and height, body mass index (BMI), neurological exam
* ECG (electrocardiography) and blood and urine tests
* Pregnancy tests for women of childbearing age
* Completion of a patient diary to record mobility and time asleep
* Parkinson's Kinetigraph (PKGTM) Data Logger: a watch-type movement recording device
* Questionnaires, rating scales and forms: quality of life, mood, memory, impulse control, mental health.
* Magnetic resonance imaging (MRI)
* Positron emission tomography scans (PET)
* Skin condition over any remaining implanted subcutaneous portion of the device.
* Skin healing after port / device removal.

For more information: https://treater.eu/clinical-study/

ELIGIBILITY:
Inclusion Criteria:

1. Completion of visit 4 (implantation of DDS) within main study HP-CD-CL-2002.
2. Patients who:

   * Discontinued main study after visit 4 of main study or discontinued extension study.
   * Received 6 doses in main study but didn't participate in extension study.
   * Received 12 doses including extension study.
3. Provision of informed consent.

Exclusion Criteria:

* None

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-09-20 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs)[safety-tolerability] | Until study completion, up to month 58
  Total number, causality and severity of adverse events at any time during the study period
Change in Electrocardiogram (ECG): Ventricular rate (bpm), [safety-tolerability] | Week 71 and Month 25
  Changes in electrical activity of heartbeat measured by electrocardiogram: Ventricular rate (bpm),
Change in Electrocardiogram (ECG): PR (pulse rate) interval, qRS duration, QT, QTc (msec) [safety-tolerability] | Week 71 and Month 25
  Changes in electrical activity of heartbeat measured by electrocardiogram: PR interval (msec), QRS duration (msec), QT (msec), QTc (msec)
Change in Beck Depression Inventory (BDI) score [safety-tolerability] | Week 71 and Month 25
  Assessment of change in depression using Beck Depression Inventory (BDI) score: Sadness: Pessimism; Past Failure; Loss of pleasure; Guilty feelings; Punishment Feelings; Self-dislike; Self-criticalness;Suicidal thoughts or wishes; Crying; Agitation; Loss of interest; Indecisiveness;Worthlessness; Loss of energy; Changes in sleeping pattern; Irritability; Changes in appetite; Concentration difficulty; Tiredness or fatique; Loss of interest in sex. Rated on a 4-point scale ranging from 0 to 3 based on severity of each item (0=low intensity; 3=highest intensity). The maximum total score is 63.
Change in Questionnaire for impulsive-compulsive disorder in Parkinson's disease rating scale (QUIP_RS) [safety-tolerability] | Week 71 and Month 25
  Assessment of changes in impulsive-compulsive disorders using QUIP_RS. Questions scored 0-4 (0=never; 4=very often) on gambling, sex, buying, eating, performing tasks/hobbies, repeating simple activities, and taking Parkinson's disease medication. Total QUIP-RS Score 0-112
  Assessment of changes in impulsive-compulsive disorders using QUIP_RS. Questions scored 0-4 (0=never; 4=very often) on gambling, sex, buying, eating, performing tasks/hobbies, repeating simple activities, and taking Parkinson's disease medication. Total QUIP-RS Score 0-112
  Assessment of changes in impulsive-compulsive disorders using QUIP_RS. Questions scored 0-4 (0=never; 4=very often) on gambling, sex, buying, eating, performing tasks/hobbies, repeating simple activities, and taking Parkinson's disease medication. Total QUIP-RS Score 0-112
Change in Montreal cognitive assessment (MoCA) [safety-tolerability] | Week 71 and Month 25
  Assessment of change in cognitive domains using MoCA test: attention and, concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total possible score is 30 points; a score of 26 or above is considered normal.
Changes in physical examination: anatomic findings [safety-tolerability] | Week 71, and Months 25, 34, 58
  Changes in anatomic findings found in physical examination of the following body systems: general inspection/upper extremities; head, eyes, ears, nose, throat, and superficial cervial lymph notes; neck, shoulders, back; chest and lungs; cardiovascular; abdomen; lower extremities
Changes in physical examination: clinical standard neurological examination | Week 71, and Months 25, 34, 58
  A clinical standard neurological examination by study investigator. Changes in motor function, sensory function, cranial nerve function (visual fields), cortical functions and reflexes are followed in the examination, scored as normal - abnormal without clinical relevance - abnormal with clinical relevance
Changes in vital signs: blood pressure [safety-tolerability] | Weeks 55, 57, 58, 75
  Changes in blood pressure during the study , measured as systolic and diastolic blood pressure (in mmHg)
Changes in vital signs: pulse rate [safety-tolerability] | Weeks 55, 57, 58, 75
  Changes in pulse rate during the study (in beats per minute)
Changes in vital signs: body temperature [safety-tolerability] | Weeks 55, 57, 58, 75
  Changes in body temperature during the study (in degrees celcius)
Changes in vital signs: body weight [safety-tolerability] | Weeks 55, 57, 58, 75
  Changes in body weight during the study (in kilograms)
Changes in vital signs: body mass index (BMI) [safety-tolerability] | Weeks 55, 57, 58, 75
  Changes in body mass index during the study (in kg/m^2)
Changes in clinical laboratory safety screen: clinical chemistry [safety-tolerability] | Weeks 53, 55, 57, 58, 71 and Months 25, 34, 58
  Changes in laboratory variables for clinical chemistry (Na, K, Urea, creatinine, creatine kinase, Ca, Bilirubin, IgG (Immunoglobulin G), Albumin, ALP(Alkaline phosphatase), ALT (Alanine transaminase), AST (Aspartate transaminase))
Changes in clinical laboratory safety screen: haematology - haemoglobin [safety-tolerability] | Weeks 53, 55, 57, 58, 71 and Months 25, 34, 58
  Changes in laboratory variables for haematology: hemoglobin (g/L). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: haematology - haematocrit [safety-tolerability] | Weeks 53, 55, 57, 58, 71 and Months 25, 34, 58
  Changes in laboratory variables for haematology: hematocrit (%, ratio of red blood cell volume to total blood volume). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: haematology - red blood cell (RBC) count [safety-tolerability] | Weeks 53, 55, 57, 58, 71 and Months 25, 34, 58
  Changes in laboratory variables for haematology: RBC count (10E12/L). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: mean cell volume (MCV) of red blood cells [safety-tolerability] | Weeks 53, 55, 57, 58, 71 and Months 25, 34, 58
  Changes in laboratory variables for haematology: MCV of red blood cells (fL). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: mean cell haemoglobin of RBC (MHC) [safety-tolerability] | Weeks 53, 55, 57, 58, 71 and Months 25, 34, 58
  Changes in laboratory variables for haematology: MCH (Mean cell hemoglobin) (pg). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: Platelet count [safety-tolerability] | Weeks 53, 55, 57, 58, 71 and Months 25, 34, 58
  Changes in laboratory variables for haematology: Platelet count (10E9/L). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: white blood call (WBC) count [safety-tolerability] | Weeks 53, 55, 57, 58, 71 and Months 25, 34, 58
  Changes in laboratory variables for haematology: Cell counts (10E9/L) for total WBC, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: activated partial thromboplastin time (aPTT) [safety-tolerability] | Weeks 53, 55, 57, 58, 71 and Months 25, 34, 58
  Changes in laboratory variables for haematology: aPTT (sec) . Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: International Normalised Ratio (INR) [safety-tolerability] | Weeks 53, 55, 57, 58, 71 and Months 25, 34, 58
  Changes in laboratory variables for haematology: INR (standardized prothrombin time) to determine the effects of oral anticoagulants on the clotting system. Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: urinanalysis [safety-tolerability] | Weeks 53, 55, 57, 58, 71 and Month 25
  Changes in laboratory variables for urinanalysis (blood/erythrocytes, glucose, ketones, leukocytes, nitrites, pH, protein) studied by dipstick and scored 0-3. Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Formation of anti-CDNF antibodies [safety-tolerability] | Weeks 58, 78 and Month 25
  Formation and change in anti-CDNF antibody concentration (in ng/ml).
Device related occurrence of adverse device effects [safety-tolerability] | Week 49 and Month 58
  Occurrence of adverse device effects (ADE) at any time of the study period, for either the whole system or the individual sub systems (guide tubes/catheters, subcutaneous components, port), serious adverse device effect (SADE) including long term effects, neurological deficit (seizures), infection (local to components, in CNS), severe skin breakdown or necrosis requiring component removal life threatening or major (requiring intervention) intracerebral haemorrhage.

SECONDARY OUTCOMES:
Change in UPDRS (Unified Parkinson's Disease Rating Scale) Part III motor score [efficacy] | Week 71 and Month 25
  Changes in severity of PD (Parkinson's disease) motor symptoms assessed by UPDRS Part III motor scores (each scored 0-4; 0=none, 4=severe): Speech; facial expression; tremor a rest; Tremor of hands; rigidity; firger taps; hand movelents; alternating movement of hands; leg agility; rising from chair; posture; gait; postural stability; body bradykinesia and hypokinesia. The total score, the sum of scores received from 27 assessments, is 0 - 108
Change in TUG (Timed Up and Go) test [efficacy] | Week 71 and Month 25
  Changes in mobility assessed by TUG test (in minutes and seconds).
Change in UPDRS Total score (Part I-IV) [efficacy] | Week 71 and Month 25
  Change in severity of PD non-motor and motor symptoms assessed by UPDRS Part I-IV total scores (Parts I, II and IV in ON-state; Part III in OFF-state): Part 1 (scored 0-16) Mentation, behaviour and mood. Part 2 (scored 0-52) Activities of daily living. Part 3 (scored 0-108) Motor examination. Part 4 (scored 0-23) Complications of therapy. The total score is 0-199 (0=totally healthy; 199=worst possible).
Change in home diary score [efficacy] | Weeks 40, 45, 49, 53, 57, 58, 61, 65, 71, and Month 25
  Change in functional status of the patient's dyskinesias assessed by home diary score for three-day period. Each half hour is scored: sleep, OFF, ON without dyskinesias, ON with non-troublesome dyskinesias, ON with troublesome dyskinesias. The total time in each state over 3 days is recorded (in hours). The total "bad time" is defined as "OFF time" and "ON time with troublesome dyskinesia". The total "good time" is defined as "ON time without dyskinesia" or "ON time with non-troublesome dyskinesia".
Change in PDQ-39 (Parkinson's Disease Questionnaire) score [efficacy] | Week 71 and Month 25
  Changes in health and daily activity assessed by a self-administered PDQ-39 questionnaire comprising of 39 questions related to eight key areas of health in Parkinson's patients: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication and bodily discomfort. Each question is evaluated on a scale of five terms "Never", "Occasionally", "Sometimes", "Often" or "Always or cannot do at all".
Change in CGI-I (Clinical Global Impression - Improvement) scale [efficacy] | Weeks 40, 45, 49, 53, 57, 58, 61, 65, 71, and Month 25
  Change in mental status as measured by CGI-I scale rated by the clinical on a seven-point scale 1-7 (1=very much improved, 4=no change, 7=very much worse).
Healing of patient skin after port removal | Month 25, 34 and 58
  Any Adverse Events (AEs) or Serious Adverse Events (SAEs) related to the skin condition once the port has been removed

OTHER OUTCOMES:
Change in DAT (dopamine transporter)-PET imaging [exploratory] | Week 63
  Change in caudate and putamen DAT availability using PET imaging
Change in daily activity measurement [exploratory] | Weeks 58, 71 and Month 25
  Change in daily activity measured by Parkinson's KinetiGraph™ (PKG™) Data Logger: dyskinesia, bradykinesia, tremor, immobility plot, fluctuation score. The PKG units are: Bradykinesia score in % from normal controls, and, Dyskinesia score in % from normal controls. The Fluctuation and Dyskinesia score (FDS) for normal controls is in the range of 7.8-12.8: a lower score indicates bradykinesia and a higher score indicates dyskinesia.

CONTACTS AND LOCATIONS:
Locations (3):
- Helsinki University Hospital, Helsinki, Finland
- Sweden (2):
  - Skåne University Hospital, Lund
  - Karolinksa University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No